CLINICAL TRIAL: NCT00504023
Title: A Pilot Study of Topical Imiquimod Therapy for the Treatment of Recurrent Extramammary Paget's Disease
Brief Title: Topical Imiquimod in Treating Patients With Recurrent Paget's Disease of the Vulva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-029; MSKCC-07029
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-02

CONDITIONS: Vulvar Cancer
Keywords: Paget disease of the vulva; recurrent vulvar cancer; stage 0 vulvar cancer; stage I vulvar cancer; stage II vulvar cancer; stage III vulvar cancer; imiquimod; 07-029
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Imiquimod; Biopsy

ARMS (1):
- imiquimod (Experimental): This is a pilot study of the use of a topical immunomodulatory agent, imiquimod, for the treatment of recurrent Extramammary Paget's disease (EMPD).
  Interventions: Drug: imiquimod; Procedure: biopsy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: imiquimod — The patient will be seen in clinic every six weeks during treatment for examination. Imiquimod cream is to be applied 3 times per week for 12 weeks.
Procedure: biopsy — Punch biopsy and photography will be performed at the baseline and 12 week time points.
Procedure: therapeutic conventional surgery — If the lesion is still present after 12 weeks of therapy, the treating physician will recommend excision of the lesion four weeks after completion of therapy (week 16).

SUMMARY:
RATIONALE: Biological therapies, such as imiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. Applying topical imiquimod to the vulva may be an effective treatment for recurrent Paget's disease.

PURPOSE: This clinical trial is studying how well topical imiquimod works in treating patients with recurrent Paget's disease of the vulva.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the clinical and histologic effects of topical imiquimod therapy on recurrent extramammary Paget's disease.

OUTLINE: This is a pilot, prospective, multicenter study.

Patients apply topical imiquimod cream to a target vulvar lesion 3 times weekly. Treatment continues for up to 12 weeks in the absence of disease progression or unacceptable toxicity. If the lesion is still present after completion of 12 weeks of imiquimod therapy, the patient undergoes surgical excision of the target lesion (and any other progressive lesions suspicious for evolving adenocarcinoma) at week 16.

Patients undergo punch biopsy and photographic assessment of a target vulvar lesion at baseline and again at 12 weeks.

After completion of imiquimod therapy or after surgical excision, patients are followed at 6 weeks and then every 3 months for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting to the Gynecology outpatient service at a participating institution who meet eligibility requirements may be included in this clinical trial. The eligibility requirements are as follows:

* Age ≥18.
* Ability to give informed consent.
* Patients must have biopsy proven recurrent extramammary Paget's disease confirmed at the participating site.

Exclusion Criteria:

* Patients with known hypersensitivity to imiquimod.
* Pregnant and nursing women are not eligible
* Patients with underlying adenocarcinoma on biopsy of lesion confirmed at the participating site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis S. Chi, MD, FACOG, FACS, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert Soslow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imiquimod
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imiquimod
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 72 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical and Histologic Remission
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 12 weeks post treatment
Measure: Number; unit: % of participants
Arm/Group | Imiquimod
Number analyzed (Participants) | 8
% of participants | 75

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Imiquimod
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imiquimod (N=8)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imiquimod (N=8)
Dry Eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain - Head/Headache (Nervous system disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT00504023/Prot_SAP_000.pdf